CLINICAL TRIAL: NCT05036902
Title: The Impact of Multimodality Treatment on Physical Functions and Quality of Life in Patients With Head and Neck Cancer: A Prospective Cohort Study
Brief Title: The Impact of Multimodality Treatment on Physical Functions and Quality of Life in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/2578
Record Dates: First submitted 2021-08-23; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral cancer (including the lip) alone, with 300.373 cases worldwide in 2012, is the predominant head and neck squamous cell carcinoma. With an incidence of 6.5 cases per 100.000, south - east asia has the highest incidence worldwide. Many of these cases do present at a locally advanced stage, which often requires combined modality treatment that includes extensive surgery to the primary site and neck and flap reconstruction. This is often followed by either adjuvant radiation or chemo-radiotherapy. This treatment can come with a significant morbidity affecting the self-care ability of the patients as well as impact the quality of life(QOL) (3,4).At the SingHealth Duke - NUS Head and Neck Centre 340 complex cases of head and neck cancer (HNC) involving flap reconstructions and extensive resections have been operated in 2014 alone. Almost all of these patients need further adjuvant treatment (radiotherapy and/or chemotherapy). Side-effects following such treatments, Significant number of patients underwent subsequent adjuvant treatment. The adjuvant treatment and surgery may render these patients weakness of the shoulder and neck muscles, numbness and reduced sensation around the neck and shoulder region and a general impact on the patient's fitness. While survival remains the most important outcome in oncologic treatment, recovery of treatment related morbidity and return to pre-treatment QOL for patients after cancer treatment is equally important.

The aims of this study is to evaluate the impact of surgical and adjuvant treatment on physical functions and QOL of the patients. By measuring the impact of extensive treatments for head and neck malignancies on the fitness and QOL of these patients, the team aims to identify the risk factors that necessitate a more aggressive rehabilitation. This is to date the first prospective study investigating the impact of multimodality treatment on fitness and QOL in HNC patients in a structured and predefined manner. Ultrasound (US) elastography will be used to assess muscle and soft tissue stiffness and elasticity and correlate these with functional outcome measurements. Elastography has been previously described as a useful tool to assess stiffness of the neck soft tissues and muscles, however no study thus far has correlated these findings with functional measurements. Hence this trial aims to establish the following:

1. Due to the limited available data: to quantify and qualify the impact of surgery as well as adjuvant treatment on the fitness, physical function of the neck and shoulder & QOL of HNC patients
2. To establish a workflow and assessment protocol for a subsequent larger prospective clinical trial
3. To identify performance markers in these patients, that allow a more targeted rehabilitation process
4. Many patients post head and neck treatment are economically compromised since they are unable to return to mainstream work and there exists a significant unemployment rate. The understanding we gain through objective analysis apart from targeted treatment for every individual patient, in the future this study hopes to address and improve the economic impact to the individual and probably reduce the health care burden.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study by recruiting patients who are admitted to NCCS for HNC surgery. It will be a pilot study targeting 10 patients to compare physical functions and QOL 1 to 2 weeks pre-surgery, 3-6 weeks post-surgery and 6 months post-surgery. The results from phase I will be used to plan the sample size for the following phase. Each visit will take approximately 4 hours.

Assessment of Physical Functions

1. Shoulder Range of Motion (ROM) and strength for both arms (1 hour):

   Routinely practiced by Physiotherapists as a part of evaluation for any patient referred for shoulder physiotherapy. These will be measured by the Dynamometer (Biodex S4 Pro) with patients in a seated position. Active and passive shoulder movements include abduction, adduction, and flexion, and extension, internal and external rotation. Strength test of the upper and lower limbs will also be performed using an isometric hand-held dynamometer. The measures will be done in the positions stated below:
   1. Bilateral knee extension at 90 degree knee flexion. Unit measure: kg
   2. Bilateral shoulder flexion at 45 degree shoulder flexion. Unit measure: kg Shoulder Pain and Disability Index (SPADI) questionnaire will also be administered to evaluate shoulder pain and impairment.
2. Point of gaze measurement (30 mins):

   A non-invasive assessment tool to assess head and neck movement. Head range of movement will be assessed pre and post treatment using a light source together with the motion capture system. Participants will be seated in the middle of the room with reflective markers placed on their head and shoulder. The participants will keep their gaze fixed on the light source and then rotate the head as far as possible without losing gaze fixation. The light source will move in different planes. This will allow the impact of surgical treatment on head and neck mobility to be assessed. Head movement, relative to the thorax will be measure in 3 dimensions. Restrictions in flexion, lateral flexion and rotation will be quantified along with angular velocity and acceleration.
3. Muscle activation patterns will also be evaluated using EMG (30 mins):

   Routinely practiced in physiotherapy.

   Sternocleidomastoid muscle:

   Sternal head and clavicular head on cervical contralateral rotation and ipsilateral cervical flexion

   Serratus anterior:

   Supine, shoulder at 90° flexion, elbow fully extended - Resistance applied into shoulder retraction

   Rhomboid major muscle:

   Prone, head rotated ipsilaterally - Scapula adducted and elevated. Elbow fully flexed, shoulder extended and adducted Resistance applied into shoulder abduction and depression

   Upper trapezius muscle:

   Scapula elevation in sitting - Resistance applied into shoulder depression and cervical spine contralateral flexion

   Middle trapezius muscle:

   Scapula elevation in sitting - Resistance applied into shoulder depression and cervical spine contralateral flexion
4. Grey-scale (B-mode) ultrasound and Shear-wave elastography imaging (1 hour) Non-invasive and of standard clinical care practice, however elastography, a non-invasive test is a new dimension to this test to assess the density and rigidity of muscles (practised in the area of breast surgery) and new application for head and neck cancer patients.

   To allow assessment of tissue stiffness via elastography the following protocol will be employed:

   Grey-scale and shear-wave ultrasound elastography will be performed at baseline (pre-op), 4-weeks and 6-months post-op. All examinations will be performed with the patient supine and neck extended; using the SuperSonic ultrasound machine (Aixplorer; SuperSonic Imagine, Aix-En-Provence, France) that equipped with a 15-MHz superficial linear transducer.

   Grey-scale (B-mode) ultrasound:

   The examination will begin with grey-scale ultrasound to assess the sternocleidomastoid (SCM, or trapezius) muscle thickness. In order to ensure consistency in image acquisition and reproducibility of the ultrasound scans at follow-up, the thickness of the SCM (or trapezius) muscle will be measured on the longitudinal plane, at the of the upper edge of the thyroid cartilage.

   The thickness measurement will be repeated once (i.e. 2 sets of thickness measurements will be obtained) and the mean values will be recorded for final analysis.

   After recording the grey-scale images, real-time shear-wave elastography will be obtained with the participants in the same position.

   Shear-wave elastography imaging:

   On longitudinal image, the SCM (or trapezius) muscle will be divided into proximal, mid and distal sections. The shear-wave elastography imaging mode will be activated.

   A rectangular acquisition box displaying the color map of differential tissue stiffness (red: stiff area; blue: soft area; and green/yellow: intermediate stiffness) will be placed in the centre of the field of view. The shear-wave velocity (in meters per second) will be measured on the longitudinal shear wave image by placing a circle ROI that covers almost the entire muscle tissues in the rectangular acquisition box.

   The shear-wave image acquisition will be repeated for mid and distal third SCM sections. 2 sets of muscle velocity (m/sec) and elasticity (kpasc) values will be recorded for each SCM section. The mean of the measurements will be used for final analysis [Note: The velocity of shear wave propagation is directly related to tissue stiffness (Velocity increases with stiffness). The entire length of SCM muscle is approximately 13-15cm. The transducer length is 5cm. The investigators divide each SCM muscle into thirds for evaluation to allow overlapping scans and maximise assessment of SCM muscle stiffness
5. Fitness

Treadmill (Modified Bruce protocol) (45 mins):

Treadmill is a time tested test as a part of cardiac and pre-anesthetic work up, however in this study the application is new perspective to assess fitness in head and neck cancer patients. The modified Bruce commenced at 2.7km/h at 0% incline for 3 minutes followed by 2.7km/h at 5% incline for 3 minutes before going to the next stage which is the real STAGE 1 of the Bruce protocol. As for estimating the VO2- there is a linear relationship between HR and VO2 peak or HRR and VO2R, provided the subjects' HR is not attenuated eg. those on beta blockers.

6-minute walk test (6MWT) (10 mins) For the 6MWT, subjects are require to walk laps of 20m at the fastest they are able to perform over the period of 6 minutes. Subjects would be allowed to stop and rest within the allocated time period.

1. Total distance. Unit measure: m
2. Predicted distance: Unit measure: %
3. Predicted VO2 max: Unit measure: mL/(kg·min) 6. Assessing sensory loss secondary to incision / flap elevation and adjuvant therapy (5 mins) Routinely practised in Neurology the application specifically for head and neck cancer patients is focused way of assessing post-operative outcome may not be routinely practiced.

Mapping Sensory Loss: Dermatomes C2 to T5 via the sharp blunt test as routinely used in neurological assessment 7. Assessment of QOL (10 mins) Has been routinely practiced in head and neck cancer and is a component of standard clinical care, however not mandatory.

QOL will be evaluated by administering the evaluated SPADI, EORTC QLQ H&N35 and EORTC QLQ C30 questionnaires, which are already used as part of the general QOL assessment of the head and neck cancer patients in the Singhealth DukeNUS Head & Neck Centre. Besides the assessments, all subjects will undergo physiotherapy intervention (approx 1 hour) immediately after surgery, once stable and allowed by the medical team all subjects will be ambulated as tolerated, as per post-operative protocol.

Two weeks after surgery or when allowed by medical team, whichever is later, the subjects will be guided to progress follow the work-out with the following routine for the period of three to six months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven cancers of the upper aero-digestive tract (oral cavity, oropharynx, nasopharynx or pharynx), skin, thyroid or salivary glands;
2. Case has been indicated for surgical treatment and following adjuvant treatment in the multidisciplinary head and neck tumour board
3. Age: 21 - 70 years
4. ECOG 0 or 1
5. Able to give informed consent

Exclusion Criteria:

1. Patients who are not able to undergo primary resection of their HNC(not fit for general anesthesia)
2. Patients with distant metastases or incurable recurrent disease
3. Patients who are currently pregnant or breastfeeding
4. Patients with a history of shoulder surgery or trauma, or any known joint pathology such as rheumatologic disorders, or prior neurological disease affecting the upper and or lower extremity such as stroke;
5. Patients who are receiving a free fibular flap as part of their reconstruction
6. Patients who are on a permanent tracheostomy e.g. after a total laryngectomy
7. Patient with ischaemic heart disease or with current beta blocker medication

Ages: 21 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients of National Cancer Centre and Singapore General Hospital that have Head and Neck Cancer
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline Shoulder Range of Motion at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  Active and passive shoulder movements include abduction, adduction, and flexion, and extension, internal and external rotation.
Change from post op 6weeks Shoulder Range of Motion at 6 months | 3-6 weeks post surgery, 6 months post surgery
  Active and passive shoulder movements include abduction, adduction, and flexion, and extension, internal and external rotation.
Change from baseline Bilateral Strength at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  Strength test of the upper and lower limbs will also be performed using an isometric hand-held dynamometer.
Change from post op 6 weeks Bilateral Strength at 6 months | 3-6 weeks post surgery, 6 months post surgery
  Strength test of the upper and lower limbs will also be performed using an isometric hand-held dynamometer.
Change from baseline Head Range of Motion at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  Head range of movement will be assessed pre and post treatment using a light source together with the motion capture system. Restrictions in flexion, lateral flexion and rotation will be quantified along with angular velocity and acceleration.
Change from post op 6 weeks Head Range of Motion at 6 months | 3-6 weeks post surgery, 6 months post surgery
  Head range of movement will be assessed pre and post treatment using a light source together with the motion capture system. Restrictions in flexion, lateral flexion and rotation will be quantified along with angular velocity and acceleration.
Change from baseline Shoulder Pain and Disability Index questionnaire at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  to evaluate shoulder pain and impairment. To answer the questions, patients place a mark on a 10cm visual analogue scale for each question. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Change from post op 6 weeks Shoulder Pain and Disability Index questionnaire at 6 months | 3-6 weeks post surgery, 6 months post surgery
  to evaluate shoulder pain and impairment. To answer the questions, patients place a mark on a 10cm visual analogue scale for each question. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Change from baseline EMG Muscle Activation Patterns at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  Sternocleidomastoid muscle, Serratus anterior, Rhomboid major muscle, Upper trapezius muscle, Middle trapezius muscle
Change from post op 6 weeks EMG Muscle Activation Patterns at 6 months | 3-6 weeks post surgery, 6 months post surgery
  Sternocleidomastoid muscle, Serratus anterior, Rhomboid major muscle, Upper trapezius muscle, Middle trapezius muscle
Change from baseline thickness of the SCM (or trapezius) muscle at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
Change from post op 6 weeks thickness of the SCM (or trapezius) muscle at 6 months | 3-6 weeks post surgery, 6 months post surgery
Change from baseline Maximum Rate of Oxygen consumption measured at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
Change from post op 6 weeks Maximum Rate of Oxygen consumption measured at 6 months | 3-6 weeks post surgery, 6 months post surgery
Change from baseline EORTC QLQ C30 (European Organisation for Research and Treatment of Cancer quality of life questionnaire) at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  Quality of Life measurement. The EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the health related quality of life (QoL) of cancer patients participating in international clinical trials. The core questionnaire, the QLQ-C30, is the product of more than a decade of collaborative research. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems
Change from post op 6 weeks EORTC QLQ C30 ((European Organisation for Research and Treatment of Cancer quality of life questionnaire) at 6 months | 3-6 weeks post surgery, 6 months post surgery
  Quality of Life measurement. The EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the health related quality of life (QoL) of cancer patients participating in international clinical trials. The core questionnaire, the QLQ-C30, is the product of more than a decade of collaborative research. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems
Change from baseline EORTC H&N35 (European Organisation for Research and Treatment of Cancer quality of life questionnaire Head and Neck Module) at 6 weeks | 1-2 weeks pre surgery, 3-6 weeks post surgery
  Quality of Life measurement. The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems (i.e. there are no function scales in which high scores would mean better functioning).
Change from post op 6 weeks EORTC H&N35 (European Organisation for Research and Treatment of Cancer quality of life questionnaire Head and Neck Module) at 6 months | 3-6 weeks post surgery, 6 months post surgery
  Quality of Life measurement. The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems (i.e. there are no function scales in which high scores would mean better functioning).

SECONDARY OUTCOMES:
Assessing sensory loss secondary to incision / flap elevation and adjuvant therapy | 1-2 weeks pre surgery, 3-6 weeks post surgery, 6 months post surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National Cancer Centre, Singapore
  - Singapore General Hospital, Singapore